CLINICAL TRIAL: NCT07124858
Title: PRODIGE 108 - COHORTE 2320 - COFRUQ Prospective National Cohort Evaluating Prognostic Factors for Efficacy of Fruquintinib Treatment in Patients With Metastatic Colorectal Cancer
Brief Title: Prospective National Cohort Evaluating Prognostic Factors for Efficacy of Fruquintinib Treatment in Patients With Metastatic Colorectal Cancer
Acronym: COFRUQ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COFRUQ COHORT; 2024-A00994-43 (Registry Identifier: ID RCB ANSM)
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Colorectal Cancer (CRC); Antineoplastic Agents, Immunological; VEGFR-TKI
Keywords: Metastatic colorectal cancer; Fruquintinib; cohort
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib (Other): Fruquintinib will be administered according to the summary of product characteristics (SmPC) : 5 mg, 21 days of treatment followed by a 7-day break until progression, unacceptable toxicity, death, or patient refusal.
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib will be administered according to the summary of product characteristics (SmPC) : 5 mg, 21 days of treatment followed by a 7-day break until progression, unacceptable toxicity, death, or patient refusal.

SUMMARY:
The main objective of this study is to identify the prognostic factors (clinico-biological) for the efficacy (overall survival) of fruquintinib in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Fruquintinib (a novel, highly selective oral tyrosine kinase inhibitor targeting VEGFR-1, -2, and -3) has demonstrated efficacy in chemotherapy-resistant metastatic colorectal cancer (mCRC) in two phase III trials, FRESCO and FRESCO-2. In France, fruquintinib has been available through compassionate use since January 16, 2024, for all patients with chemotherapy-refractory mCRC, and its reimbursement is expected in the coming months. However, limited real-world data are currently available regarding the use of this new treatment and the identification of predictive factors of its efficacy, both clinically and biologically.

Moreover, there is a significant lack of information concerning older patients (≥70 years), who are often underrepresented in registration trials. This cohort will therefore provide a unique opportunity to gather specific data in elderly patients, including the integration of geriatric assessment parameters.

The main objectives of this cohort will be to validate, in routine clinical practice, the survival and safety outcomes observed in the FRESCO-2 trial, and to identify clinical and biological prognostic and predictive factors of survival in patients treated with fruquintinib.

As such, the COFRUQ cohort could help identify patients who derive the greatest survival benefit from fruquintinib and thereby contribute to optimizing their therapeutic pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over.
* Histologically confirmed colorectal adenocarcinoma with locally advanced disease and/or unresectable metastasis(es) receiving treatment with fruquintinib under i) compassionate/early access and ii) marketing authorisation and reimbursement in France.
* Obtain informed consent from the patient for the clinical-biological cohort.
* Agreement to take biological samples of ctDNA and send tumour blocks (patient participation in the pharmacokinetic study remains optional).

Exclusion Criteria:

* Patient with another concurrent cancer at the time of diagnosis, requiring systemic treatment or influencing prognosis (in the opinion of the centre's medical team).
* Contraindication due to psychological or social reasons that may hinder follow-up (cognitive deficit, psychological disorders incompatible with obtaining consent; inability to be followed in the same centre throughout the follow-up period for geographical reasons).
* Pregnant or breast-feeding women.
* Patients under court protection or subject to a protective measure (patient under guardianship or curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 1 year after treatment start
  OS is defined as the time interval (months) between the date of initiation of treatment with fruquintinib and the date of death (from any cause).

SECONDARY OUTCOMES:
progression free survival | up to 1 year after treatment start
  Time (months) from initiation of treatment with fruquintinib to radiological and/or clinical tumour progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (83):
- France (83):
  - Poitiers CHU, Poitiers, France
  - Centre Hospitalier, Albi
  - CHU, Amiens
  - Clinique de L Europe, Amiens
  - Centre Hospitalier, Annecy
  - Centre Hospitalier, Aurillac
  - Centre Hospitalier, Bayeux
  - Centre Hospitalier, Bayonne
  - Centre Hospitalier, Beauvais
  - CHU, Besançon
  - Centre Hospitalier Bethune Beuvry, Beuvry
  - Centre Pierre Curie, Beuvry
  - Clinique Tivoli, Bordeaux
  - Polynclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHU, Brest
  - CHU, Caen
  - Centre Hospitalier, Calais
  - Infirmerie Protestante, Caluire-et-Cuire
  - Clinique Sainte Marie, Chalon-sur-Saône
  - ROC37, Chambray-lès-Tours
  - Centre Hospitalier, Chartres
  - Centre Hospitalier, Cholet
  - Clinique Sainte Come, Compiègne
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Clinique Branche - Clinique Flandres, Coudekerque-Branche
  - Centre Hospitalier Henri Mondor, Créteil
  - Centre Leonard de Vinci, Dechy
  - Chu Francois Mitterand, Dijon
  - Institut de Cancerologie de Bourgogne, Dijon
  - Hopital Prive Forcilles, Férolles-Attilly
  - Centre Hospitalier, Flers
  - CHI, Fréjus
  - Groupe Hospitalier Mutualiste, Grenoble
  - Polyclinique de Blois, La Chaussée-Saint-Victor
  - Clinique Sainte Clothilde, La Réunion
  - Centre Hospitalier de Vendee, La Roche-sur-Yon
  - Hopital Prive de L Estuaire, Le Havre
  - Centre Hospitalier, Le Puy-en-Velay
  - Centre Hospitalier, Lens
  - CHU, Lille
  - CHU, Limoges
  - Groupement Hospitalier Bretagne Sud, Lorient
  - Clinique Jean Mermoz, Lyon
  - Hopital Europeen, Marseille
  - Hopital Saint Joseph, Marseille
  - La Timone, Marseille
  - Clinique Gray, Maubeuge
  - Ch Du Mittan, Montbéliard
  - Institut de Cancerologie de Lorraine, Nancy
  - Hopital Prive Confluent, Nantes
  - Clinique Ambroise Pare Hartmann, Neuilly
  - Hopital Americain, Neuilly-sur-Seine
  - Centre Hospitalier, Niort
  - CH de la source, Orléans
  - BICHAT, Paris
  - COCHIN, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hopital Avicenne, Paris
  - Hopital Saint Louis, Paris
  - La Pitie Salepetriere, Paris
  - Saint Antoine, Paris
  - Centre Hospitalier, Pau
  - Hopital Instruction Des Armees, Percy
  - Centre Hospitalier, Perpignan
  - CHU, Pessac
  - Lyon Sud, Pierre-Bénite
  - Centre Cario, Plérin
  - CHU, Poitiers
  - CHU, Reims
  - CHU, Rennes
  - CHU, Rouen
  - Centre Hospitalier, Saint-Denis
  - Centre Hospitalier, Soissons
  - Centre Hospitalier, St-Malo
  - Clinique Sainte Anne, Strasbourg
  - Centre Hospitalier, Thonon-les-Bains
  - Chu Rangueil, Toulouse
  - CHU, Tours
  - Hopital Prive Drome Ardeche, Valence
  - CHU, Vandœuvre-lès-Nancy
  - Centre Hospitalier, Versailles
  - Hopital Nord Ouest, Villefranche-sur-Saône
  - Medipole Hopital Mutualiste, Villeurbanne